CLINICAL TRIAL: NCT04608799
Title: Director of Child Neurology, Department of Pediatrics, National Taiwan University Hospital
Brief Title: The Efficacy of Fycompa (Perampanel) in Children With Epilepsy
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201802018RIND
Record Dates: First submitted 2020-10-20; First posted 2020-10-29 (Actual); Last update posted 2020-10-29 (Actual); Status verified 2020-10

CONDITIONS: Neurologic Disorder
MeSH Terms: conditions — Nervous System Diseases | interventions — perampanel

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Perampanel — Efficacy of epilepsy drugs

SUMMARY:
Fycompa (Perampanel), a new anti-epileptic drug that uses a new mechanism-AMPA receptor antagonist. Its initial indication is for local or generalized epilepsy in children and adults over 12 years old, but its effectiveness in the treatment of epilepsy in children At present, more evidence is still needed. We will study the effectiveness of Fycompa (Perampanel) in the treatment of epilepsy in children under the age of 18. It is expected that the clinical use of Fycompa (Parampanel) in Taiwan will be able to analyze and study the effectiveness of the clinical use of Fycompa (Parampanel) in the treatment of epilepsy in children, and compare it with foreign reports.

ELIGIBILITY:
Inclusion Criteria:

* Patients under 18 years of age suffering from epilepsy
* Patients who are taking Paraampanel

Exclusion Criteria:

* Patients who are not in the above age groups and who are not using parampanel

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients suffering from epilepsy
Sampling Method: Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-03-19 (Actual); Study Completion 2020-03-19 (Actual)

PRIMARY OUTCOMES:
The efficacy of perampanel in young children with drug-resistant epilepsy | 17 years
  Because the current clinical research data on the use of Fycompa (perampanel) in children for the treatment of epilepsy is still insufficient, the purpose of this research is to review the efficacy of this drug in the treatment of children with epilepsy in our hospital in the past, so as to facilitate the future clinical treatment of children with epilepsy. Children have the possibility of therapeutic reference.

CONTACTS AND LOCATIONS:
Overall Officials: WangTso Lee, MD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No